CLINICAL TRIAL: NCT05304923
Title: Supraglottic Jet Oxygenation and Ventilation (SJOV) for Hypoxemia During Deep Sedation for Gastrointestinal Endoscopy at High-altitude
Brief Title: Supraglottic Jet Oxygenation and Ventilation for Gastrointestinal Endoscopy at High-altitude
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Tibet Autonomous Region People's Hospital (Other)
Responsible Party: Principal Investigator, Yi Feng, MD, Chair of Department of Anesthesiology, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SJOVGETBHP
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Hypoxia; High Altitude
MeSH Terms: conditions — Hypoxia; Altitude Sickness | interventions — Ventilation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supraglottic jet oxygenation and ventilation (Experimental): Supraglottic jet oxygenation and ventilation is conducted for the participants during sedation.
  Interventions: Procedure: Supraglottic jet oxygenation and ventilation
- nasal cannula oxygen supply (Placebo Comparator): Oxygen supplementation is delivered via a nasal cannula to the participants during sedation.
  Interventions: Procedure: Nasal cannula oxygen supply

INTERVENTIONS:
Procedure: Supraglottic jet oxygenation and ventilation — Supraglottic jet oxygenation and ventilation is conducted using a Wei nasal jet tube (WNJ, Well Lead Medical Co. Ltd, Guangzhou, China) which is connected to a manual jet ventilator (Well Lead Medical Co. Ltd, Guangzhou, China) via its jet port. The initial settings of SJOV are: driving pressure (DP) 15psi, respiratory rate (RR) 20 bpm, inspiratory-to-expiratory (I/E) ratio 1:2, and gas supply 100% oxygen.
  Arms: Supraglottic jet oxygenation and ventilation
Procedure: Nasal cannula oxygen supply — Oxygen supplementation at 2 liters min-1 is delivered via a nasal cannula
  Arms: nasal cannula oxygen supply

SUMMARY:
This study aims to determine whether the use of SOJV could reduce the rate of hypoxia during gastrointestinal endoscopic procedures in deeply sedated patients sedated at high altitude comparing to the supplemental oxygen administration via nasal cannula.

DETAILED DESCRIPTION:
The participants will be randomly allocated to either SJOV or nasal cannula oxygen supply in a 1:1 ratio using block randomization with variable block sizes of four or six randomized. In the nasal cannula oxygen supply group, oxygen supplementation at 2 liters min-1 is delivered via a nasal cannula. In the SJOV group, SJOV is conducted using a Wei nasal jet tube (WNJ, Well Lead Medical Co. Ltd, Guangzhou, China) which is connected to a manual jet ventilator (Well Lead Medical Co. Ltd, Guangzhou, China) via its jet port.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older;
2. underwent routine gastrointestinal endoscopy under procedural sedation;
3. consented to participate in this trial. -

Exclusion Criteria:

1. infection of the upper airway;
2. anatomical abnormalities of the face, nose, and upper airway;
3. coagulopathies;
4. anticipated or known difficult airway;
5. known allergy against propofol, soybeans, and egg;
6. absence from the high-altitude environment during the past 3 months. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-04-21 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Hypoxia during sedation | During sedation procedure
  An SPO2 of 75 - 89% for < 60 s

SECONDARY OUTCOMES:
respiratory-related complications | During sedation procedure
  pulmonary aspiration, respiratory depression (SPO2 = 90-95%) and severe hypoxia (SPO2 < 75% or < 90% for > 60s)
cardiovascular-related complications | During sedation procedure
  hypotension (systolic blood pressure < 90 mmHg), hypertension (systolic blood pressure > 160 mmHg), bradycardia (heart rate < 50 beats/min), tachycardia (heart rate > 120 beats/min)
fatal complications | from sedation initiation to 20 min after patients are awake
  severe anaphylactic reactions, myocardial infarction, cardiac arrest and death

OTHER OUTCOMES:
Adverse events related to Supraglottic Jet Oxygenation and Ventilation | 20 min after patients are awake
  pharyngalgia, xerostomia, nasal bleeding, and barotrauma

CONTACTS AND LOCATIONS:
Overall Officials: Yi Feng, Principal Investigator — Peking University People's Hospital
Locations (1):
- Tibet autonomous region people's hospital, Lhasa, Tibet, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jiang B, Li Y, Ciren D, Dawa O, Feng Y, Laba C. Supraglottic jet oxygenation and ventilation decreased hypoxemia during gastrointestinal endoscopy under deep sedation at high altitudes: a randomized clinical trial. BMC Anesthesiol. 2022 Nov 14;22(1):348. doi: 10.1186/s12871-022-01902-3. PMID 36376852